CLINICAL TRIAL: NCT00692263
Title: The Effect of Escitalopram on the Pharmacokinetics and Pharmacodynamics of Tramadol in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Professor, M.D. Kim Brosen, Institute of Pyblic Health, Clinical Pharmacology, University of Soutern Denmark
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AKF-372; EudraCT: 2007-004470-10
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Last update posted 2008-09-10 (Estimated); Status verified 2008-09

CONDITIONS: Healthy
Keywords: Healthy subjects
MeSH Terms: interventions — Escitalopram; Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): Escitalopram - tramadol
  Interventions: Drug: escitalopram and tramadol
- B (Experimental): Placebo - tramadol
  Interventions: Drug: placebo and tramadol
- C (Experimental): placebo - placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: escitalopram and tramadol — 10 mg escitalopram for 3 days 20 mg escitalopram for 6 days 150 mg tramadol as a single dose on day 9
  Other Names: Lexapro; Ultram
  Arms: A
Drug: placebo — placebo identical for 10 mg/ 20 mg escitalopram and 150 mg tramadol
  Arms: C
Drug: placebo and tramadol — 9 days of placebo equivalent to 10 / 20 mg escitalopram, one single dose of 150 mg tramadol on day 9
  Other Names: placebo; Ultram
  Arms: B

SUMMARY:
Escitalopram will be given to a panel of 16 healthy subject for 9 days. On the ninth day a single dose of tramadol is administered to the subjects and pharmacokinetic(PK) and pharmacodynamic(PD) measurements are done for the next 24 hours.

It is stated that escitalopram is only a weak inhibitor of CYP2D6 and therefore no effect is seen in Pk or PK of tramadol

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age: 18 - 45 years
* CYP2D6 phenotyped as extensive metabolizer
* CYP2C19 phenotyped as extensive metabolizer

Exclusion Criteria:

* Alcohol or drug abuse

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
AUC of (+)-M1 metabolite of tramadol | 24 hours

SECONDARY OUTCOMES:
Dynamic pupillometry | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kim Brosen, MD, D.Sc, Study Chair — Institute of Public Healht, Clinical Pharmacology, University of Southern Denmark
Locations (1):
- Institute of Public Health, Clinical Pharmacology, University of Southern Denmark, Odense, Denmark